CLINICAL TRIAL: NCT01682044
Title: Phase II Clinical Trial of Rituximab in Combination With Pegfilgrastim in Patients With Indolent B-Cell (CD-20-Positive) Lymphoma
Brief Title: Pegfilgrastim and Rituximab in Treating Patients With Untreated, Relapsed, or Refractory Follicular Lymphoma, Small Lymphocytic Lymphoma, or Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 83106; NCI-2011-00134 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00524628 (obsolete NCT alias)
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pegfilgrastim; Rituximab; Flow Cytometry; Biopsy; Immunohistochemistry; Blotting, Western

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (colony-stimulating factor and monoclonal antibody) (Experimental): Patients receive pegfilgrastim SC followed by rituximab IV 3 days later in weeks 1, 3, 5, 7, 15, 23, 31, and 39. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: pegfilgrastim; Biological: rituximab; Other: flow cytometry; Procedure: biopsy; Other: immunohistochemistry staining method; Genetic: western blotting

INTERVENTIONS:
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: flow cytometry — Correlative studies
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot

SUMMARY:
This phase II trial studies the side effects and how well giving pegfilgrastim together with rituximab works in treating patients with untreated, relapsed, or refractory follicular lymphoma, small lymphocytic lymphoma (SLL), or marginal zone lymphoma (MZL). Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of therapy. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or tumor cancer-killing substances to them. Giving pegfilgrastim together with rituximab may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of Pegfilgrastim in combination with rituximab in patients with untreated or relapsed/refractory follicular, SLL or MZL.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy (including overall response rate and durability of objective responses) of Pegfilgrastim in combination with rituximab in patients with untreated or relapsed/refractory follicular, SLL or MZL.

II. To evaluate functional and phenotypic characteristics of host neutrophils undergoing treatment with Pegfilgrastim and rituximab.

III. To evaluate changes in cluster of differentiation (CD)20 antigen expression and density of expression in patients receiving Pegfilgrastim and rituximab.

IV. To evaluate changes in serum levels of tumor necrosis factor (TNF), interferon alpha (INFalpha) and free radical levels in patients undergoing treatment with Pegfilgrastim and rituximab.

OUTLINE:

Patients receive pegfilgrastim subcutaneously (SC) followed by rituximab intravenously (IV) 3 days later in weeks 1, 3, 5, 7, 15, 23, 31, and 39. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 1 year, every 6 months for 2 years, and then yearly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Untreated or relapsed/refractory follicular, SLL or MZL (i.e. no limit to number of prior treatments as long as patients meet other study criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Measurable tumor size (at least one node measuring 4 cm^2 in bidimensional measurement)
* Expected survival of > 6 months
* Prior rituximab or other monoclonal immunotherapy permitted and eligible for rituximab monotherapy
* Full recovery from any significant toxicity associated with prior surgery, radiation therapy, chemotherapy, or immunotherapy
* Absolute neutrophil count > 1.0 x 10^9/L
* Platelets > 50 x 10^9/L
* Patients may receive erythropoietin growth factors to maintain adequate hemoglobin levels (>= 8.0 mg/dl)
* Creatinine < 1.5 x upper normal levels (UNL)
* Total bilirubin < 1.5 mg/dL (> 25.65 umol/L)
* Aspartate aminotransferase < 5 x UNL
* Alkaline phosphatase < 5 x UNL
* Informed consent approved in institutional review board (lRB)
* CD20+ B-cell lymphoma

Exclusion Criteria:

* Prior history of human immunodeficiency virus (HIV)-positivity (routine HIV testing is required pretreatment)
* Serious non-malignant disease (e.g. active uncontrolled bacterial, viral, or fungal infections) or other conditions which, in the opinion of the principal investigator would compromise other protocol objectives
* Presence of central nervous system (CNS) lymphoma
* Chemotherapy within 4 weeks of the first scheduled study treatment
* Another primary malignancy (other than squamous or basal cell carcinoma of the skin or in-situ carcinoma of the cervix) for which the patient has not been disease-free for at least five years
* Major surgery, other than diagnostic surgery, within four weeks
* Patients with non-Hodgkin lymphoma (NHL) other than relapsed/refractory follicular, MZL or SLL
* Patients must not have a history of cardiac disease, defined as New York Heart Association Class II or greater or clinical evidence of congestive heart failure
* Concurrent use of other investigational agents
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator
* Known hypersensitivity to any recombinant E coli-derived product, murine proteins, or any components of the study medications
* Concerns for the subject's compliance with the protocol
* Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g. myelodysplastic syndromes, acute or chronic myelogenous leukemia)
* Patient is currently enrolled in, or has not yet completed at least 30 days since ending another investigational device or drug trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04-17; Primary Completion 2013-11-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Hernandez-ILizaliturri, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Started | 20
Completed | 16
Not Completed | 4
Not completed — Death | 1
Not completed — Progression | 3

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Frequency of Adverse Events, Graded According to NCI CTCAE v3.0. Grade 1: Mild AE; Grade 2: Moderate AE; Grade 3: Severe AE; Grade 4: Life-threatening or disabling AE; Grade 5: Death related to AE
Time Frame: Up to 90 days after the last dose of study drugs
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
Participants
  Grade 1 | 3
  Grade 2 | 9
  Grade 3 | 6
  Grade 4 | 1
  Grade 5 | 1

2. Secondary Outcome: Overall Response Rate
Description: Overall Response is defined as Complete Response: During observation, no disease is apparent, including measurable and non-measurable disease, and no evidence of disease is observed for at least 28 days, as confirmed by a second assessment following the original observation of no disease; and Partial Response: A 50% or greater decrease from baseline in the sum of the products of the longest perpendicular diameters of all the measured lesions is noted for at least 28 days as confirmed by a second assessment following the observation of the 50% or greater decrease, and no appearance of new lesions is noted.
Time Frame: Up to 43 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
percentage of participants | 60 [38.7 to 78.1]

3. Secondary Outcome: Percent Change in Functional and Phenotypic Characteristics of Host Neutrophils From Baseline
Description: Mean percent change in CD11b level from baseline at each visit
Time Frame: Baseline and weeks 1, 3, 5, 7, 15, 23, 31, and 39
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
percent change
  week 1 | -20.2 (34.0)
  week 3 | -35.5 (28.3)
  week 5 | -24.7 (117.7)
  week 7 | -56.8 (27.4)
  week 15 | -23.8 (40.1)
  week 23 | -19.7 (35.7)
  week 31 | -18.7 (47.0)
  week 39 | -10.1 (42.7)

4. Secondary Outcome: Percent Change in CD20 Antigen Expression and Density of Expression
Description: Percent change in CD20 antigen expression and density of expression
Time Frame: At 4 years
Population: Samples tissues were not large enough to perform analysis. No participants were analyze.
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 0

5. Secondary Outcome: Percent Change in Serum Levels of Tumor Necrosis Factor (TNF) From Baseline
Description: Mean percent change in TNF level from baseline at each visit.
Time Frame: Baseline and weeks 1, 3, 5, 7, 15, 23, 31, and 39
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
percent change
  week 1 | 51.5 (65.1)
  week 3 | 14.5 (47.7)
  week 5 | 11.2 (50.1)
  week 7 | 8.3 (34.2)
  week 15 | 42.7 (76.4)
  week 23 | 27.2 (80.6)
  week 31 | 45.6 (100.5)
  week 39 | 50.2 (110.6)

6. Secondary Outcome: Percent Change in Serum Levels of Interferon Alpha (INF) From Baseline
Description: Mean percent change in INF level from baseline.
Time Frame: Baseline and weeks 1, 3, 5, 7, 15, 23, 31, and 39
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
percent change
  week 1 | -18.8 (33.2)
  week 3 | -27.8 (42.9)
  week 5 | 48.1 (124.6)
  week 7 | 8.0 (71.4)
  week 15 | 1.5 (78.6)
  week 23 | -14.1 (43.9)
  week 31 | -33.0 (49.5)
  week 39 | -7.5 (45.1)

7. Secondary Outcome: Percent Change in Serum Levels of Free Radical Levels (MFI) From Baseline
Description: Mean percent change in MFI level from baseline.
Time Frame: Baseline and weeks 1, 3, 5, 7, 15, 23, 31, and 39
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Number analyzed (Participants) | 20
percent change
  week 1 | -32.0 (66.8)
  week 3 | -22.4 (71.0)
  week 5 | -45.4 (66.5)
  week 7 | -20.4 (89.9)
  week 15 | -5.8 (137.6)
  week 23 | 0.4 (219.1)
  week 31 | 295.8 (996.1)
  week 39 | 16.0 (285.6)

ADVERSE EVENTS:
Arm/Group | Treatment (Colony-stimulating Factor and Monoclonal Antibody)
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Colony-stimulating Factor and Monoclonal Antibody) (N=20)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Colony-stimulating Factor and Monoclonal Antibody) (N=20)
Anaemia (Blood and lymphatic system disorders) | 11 (15)
Leukopenia (Blood and lymphatic system disorders) | 4 (11)
Lymphopenia (Blood and lymphatic system disorders) | 8 (25)
Neutropenia (Blood and lymphatic system disorders) | 2 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (14)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (10)
Vomiting (Gastrointestinal disorders) | 4 (5)
Asthenia (General disorders) | 2 (2)
Chills (General disorders) | 6 (8)
Discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Infusion site pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 2 (2)
Sensation of foreign body (General disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 6 (6)
Cellulitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood albumin (Investigations) | 1 (1)
Blood alkaline phosphatase (Investigations) | 15 (52)
Blood alkaline phosphatase increased (Investigations) | 3 (5)
Blood creatine (Investigations) | 1 (1)
Blood creatinine (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (3)
Blood glucose (Investigations) | 1 (1)
Blood glucose decreased (Investigations) | 1 (2)
Blood potassium decreased (Investigations) | 1 (2)
Blood sodium (Investigations) | 2 (2)
Blood sodium decreased (Investigations) | 1 (1)
Blood sodium increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 4 (10)
Body temperature increased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 3 (3)
Weight increased (Investigations) | 1 (1)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (17)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation mucosal (Nervous system disorders) | 1 (3)
Dizziness (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 4 (5)
Anorexia nervosa (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Bladder discomfort (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Pallor (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT01682044/Prot_SAP_000.pdf